CLINICAL TRIAL: NCT04077164
Title: Need Supportive Interpersonal Behaviors and Physical Activity in the Context of Couples and Chronic Pain
Brief Title: Chronic Pain, Couples, & Physical Activity
Status: Terminated | Type: Observational
Why Stopped: Resources not available.
Sponsor: Illinois Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#2019-027
Record Dates: First submitted 2019-08-05; First posted 2019-09-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain; Fibromyalgia; Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis; Ankylosing Spondylitis; Rheumatoid Arthritis; Chronic Low-back Pain; Chronic Shoulder Pain
Keywords: Couples; Relationships; Physical Activity
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis; Spondylitis, Ankylosing; Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Chronic Pain: Individuals who identify as having a chronic musculoskeletal pain condition.
  Interventions: Other: No intervention, observational only.
- Partners: Partners (e.g., life partner, spouse, or significant other) of the individual with the chronic musculoskeletal pain condition.
  Interventions: Other: No intervention, observational only.

INTERVENTIONS:
Other: No intervention, observational only. — No intervention, this study will use self-report information regarding health, social, and behavioral factors for each member of the couple.

SUMMARY:
Chronic pain affects more than 50 million adults in the United States and is estimated to cost the nation more than $560 billion dollars each year. Regular physical activity is widely recognized as essential for maintaining health for all individuals, but is particularly important for individuals with chronic pain (ICPs) as physical activity can prevent further deconditioning and may even improve pain outcomes. Previous literature has shown that certain categories of partner behaviors (e.g., solicitous, punishing, distracting) are associated with different health outcomes for ICPs, and recently researchers have begun examining partner behaviors through the lens of Self-Determination Theory, specifically looking at the effects of autonomy support from a spouse on physical activity among ICPs. Partner autonomy support has been positively associated with physical activity levels and better health outcomes, but no studies to date have explored what factors predict whether or not a partner will use an autonomy supportive interpersonal style (as opposed to a controlling interpersonal style) with the ICP.

Similarly, more research is needed on the mechanisms by which autonomy support promotes positive outcomes for ICPs. Though receiving autonomy support has been linked to increased physical activity and improved mental health, no studies have yet tested the full Self-Determination Theory model as one possible explanation of the link between this form of partner support and desirable health outcomes. In particular, it is important to understand the ICP's perspective on how partner autonomy support influences need satisfaction and autonomous motivation as possible mediators between autonomy support and ICP physical activity. Furthermore, little research has explored other need supportive behaviors or their need frustrating counterparts. The current study will not only provide greater understanding of autonomy support, but will also expand the literature regarding these other need supportive and need thwarting behaviors.

Lastly, given the value of need supportive behaviors from one's partner, it is essential to evaluate how partner perceptions of those need supportive behaviors align with ICP's perceptions of those behaviors. Any need support a partner provides is likely moderated by the ICP's perception of that support.

DETAILED DESCRIPTION:
Chronic pain affects more than 50 million adults in the United States and is estimated to cost the nation more than $560 billion dollars each year. Regular physical activity is widely recognized as essential for maintaining health for all individuals, but is particularly important for individuals with chronic pain (ICPs) as physical activity can prevent further deconditioning and may even improve pain outcomes. Previous literature has shown that certain categories of partner behaviors (e.g., solicitous, punishing, distracting) are associated with different health outcomes for ICPs, and recently researchers have begun examining partner behaviors through the lens of Self-Determination Theory, specifically looking at the effects of autonomy support from a spouse on physical activity among ICPs. Partner autonomy support has been positively associated with physical activity levels and better health outcomes, but no studies to date have explored what factors predict whether or not a partner will use an autonomy supportive interpersonal style (as opposed to a controlling interpersonal style) with the ICP.

Similarly, more research is needed on the mechanisms by which autonomy support promotes positive outcomes for ICPs. Though receiving autonomy support has been linked to increased physical activity and improved mental health, no studies have yet tested the full Self-Determination Theory model as one possible explanation of the link between this form of partner support and desirable health outcomes. In particular, it is important to understand the ICP's perspective on how partner autonomy support influences need satisfaction and autonomous motivation as possible mediators between autonomy support and ICP physical activity. Furthermore, little research has explored other need supportive behaviors or their need frustrating counterparts. The current study will not only provide greater understanding of autonomy support, but will also expand the literature regarding these other need supportive and need thwarting behaviors.

Lastly, given the value of need supportive behaviors from one's partner, it is essential to evaluate how partner perceptions of those need supportive behaviors align with ICP's perceptions of those behaviors. Any need support a partner provides is likely moderated by the ICP's perception of that support.

Self-determination theory (SDT) posits that contextual, perceptual, and individual factors may influence how much an individual uses an autonomy supportive interpersonal style through the mediators of basic psychological need satisfaction and on autonomous motivation.

The present study used path analysis to test a SDT model of the relationships between a contextual factor (autonomy support from health care provider), a perceptual factor (partner's perception of ICP motivation for physical activity), an individual factor (partner catastrophizing about ICP's pain), and the sequential mediators of relationship need satisfaction and autonomous motivation with respect to the dependent variable of partner's use of an autonomy supportive interpersonal style.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a relationship for at least 1 year or more.
* Both individuals in the relationship are 18 years or older.
* One individual in the relationship identifies as having a chronic musculoskeletal pain condition.

Exclusion Criteria:

* One or both individuals are 17 years old or younger.
* Neither individual identifies as having a chronic musculoskeletal pain condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will survey couples where one individual has a chronic musculoskeletal pain condition. Couples will be recruited from convenience samples via community organizations, support groups for individuals with chronic pain, and pain management service providers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity as Assessed by the Physical Activity Scale for Individuals with Physical Disabilities [PASIPD] | Past seven days (Prior to when participant takes cross-sectional survey.)
  This 13-item scale measures physical activity among individuals with physical disabilities. Respondents report approximately how much time they engage in 1) home repair and lawn and garden work, 2) housework, 3) vigorous sport and recreation, 4) moderate sport and recreation, and 5) occupation and transportation. Respondents answer on a 4-point Likert scale, with responses ranging from 1 (Never) to 4 (Often) or from 1 (Less than 1 hr) to 4 (More than 4hr). Items 2-13 are used to calculate the total score; the average hours per day in an activity are multiplied by a value of metabolic equivalents (METs, provided with the PASIPD scale), these values are then summed to calculate the total MET hour/day.
Use of Need Supportive Interpersonal Behaviors as Assessed by "Interpersonal Behaviors Questionnaire" (Self-report Version) [IBQ-Self] | Up to 2 weeks. Participant will answer while completing cross-sectional survey, for most this is less than 30 minutes, however, participants have up to 2 weeks to complete survey. Participant responds regarding how they usually interact with partner.
  The IBQ-Self is a 24-item self-report scale that measures how much an individual engages with others via behaviors that either support or thwart basic psychological needs (autonomy, competence, & relatedness). There are six subscales, each consists of four items, which are summed to provide a subscore, ranging from 4 to 28. Higher scores for a subscale indicate that an individual perceives they use those particular behaviors more frequently. Higher scores for autonomy support, competence support, and relatedness support are considered desirable, while lower scores for autonomy thwarting, competence thwarting, and relatedness thwarting are also viewed as more adaptive. Cronbach's alphas for the six subscales indicate acceptable reliability (αs = 0.77 to 0.82).

SECONDARY OUTCOMES:
Frequency of Depressive Symptoms as Assessed by Center for Epidemiologic Studies Depression Scale (CES-D-10) | Past week (Prior to when participant takes cross-sectional survey.)
  The CES-D-10 is a self-report measure that assesses depressive symptomatology. Respondents rate items on a 4-point Likert scale describing how often the participant felt or behaved in a certain way during the past week. The responses range from 0 "Rarely or none of the time (less than 1 day)" to 3 "Most or all of the time (5-7 days)." A total score on the CES-D-10 is yielded by summing the scores for all items, and may range from 0 to 30. A score of 10 or greater is used as a screening cutoff to indicate the presence of depression. Lower scores indicate fewer depressive symptoms and are considered desirable. The scale has good reliability, a = 0.89.
Frequency of Anxiety Symptoms as Assessed by GAD-7 | Past 2 weeks (Prior to when participant takes cross-sectional survey.)
  The GAD-7 is a 7-item self-report measure that assesses symptomatology consistent with generalized anxiety disorder. Each item is rated on a 4-point Likert scale describing how often the participant has experienced possible symptoms. The responses range from 0 "Not at all" to 3 "Nearly every day." Total scores are calculated for the GAD-7 by summing all the items, and may range from 0 to 21. Lower scores indicate fewer anxiety symptoms and are indicative of greater wellbeing. A cut point score of 10 or higher has been shown to have good specificity (89%) and sensitivity (82%) for identifying individuals with and without generalized anxiety disorder. The GAD-7 has demonstrated good internal consistency, with Cronbach's alpha at 0.92.
Use of Need Supportive Interpersonal Behaviors as Assessed by Interpersonal Behaviors Questionnaire (Other-report Version) [IBQ-Other] | Up to 2 weeks. Participant will answer while completing cross-sectional survey, for most this is less than 30 minutes, however, participants have up to 2 weeks to complete survey. Participant responds regarding how partner typically interacts with them.
  The IBQ-Other is a 24-item self-report scale that measures how an individual perceives others' interactions with them in terms of supporting or thwarting the respondent's basic psychological needs (autonomy, competence & relatedness). There are six subscales, each consists of four items, which are summed to provide a subscore ranging from 4 to 28. Higher scores for a subscale indicate that an individual perceives that people they interact with use those particular behaviors more frequently. Higher scores for autonomy support, competence support, relatedness support, and lower scores for autonomy thwarting, competence thwarting, and relatedness thwarting are considered desirable. Cronbach's alphas for the six subscales indicate acceptable reliability (αs = 0.75 to 0.89).

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Jeong Lee, PhD, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently there are no plans to share IPD with other researchers.

REFERENCES:
- [Background] Rocchi, M., Pelletier, L., Cheung, S., Baxter, D., & Beaudry, S. (2017). Assessing need-supportive and need-thwarting interpersonal behaviours: The Interpersonal Behaviours Questionnaire (IBQ). Personality and Individual Differences, 104, 423-433.
- [Background] Washburn RA, Zhu W, McAuley E, Frogley M, Figoni SF. The physical activity scale for individuals with physical disabilities: development and evaluation. Arch Phys Med Rehabil. 2002 Feb;83(2):193-200. doi: 10.1053/apmr.2002.27467. PMID 11833022
- [Background] Rocchi M, Pelletier LG. The Antecedents of Coaches' Interpersonal Behaviors: The Role of the Coaching Context, Coaches' Psychological Needs, and Coaches' Motivation. J Sport Exerc Psychol. 2017 Oct 1;39(5):366-378. doi: 10.1123/jsep.2016-0267. Epub 2017 Dec 18. PMID 29251089
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] Markland, D., & Tobin, V. (2004). A modification to the behavioural regulation in exercise questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology, 26(2), 191-196.
- [Background] La Guardia JG, Ryan RM, Couchman CE, Deci EL. Within-person variation in security of attachment: a self-determination theory perspective on attachment, need fulfillment, and well-being. J Pers Soc Psychol. 2000 Sep;79(3):367-84. doi: 10.1037//0022-3514.79.3.367. PMID 10981840
- [Background] Sabourin S, Valois P, Lussier Y. Development and validation of a brief version of the dyadic adjustment scale with a nonparametric item analysis model. Psychol Assess. 2005 Mar;17(1):15-27. doi: 10.1037/1040-3590.17.1.15. PMID 15769225
- [Background] Kerns RD, Turk DC, Rudy TE. The West Haven-Yale Multidimensional Pain Inventory (WHYMPI). Pain. 1985 Dec;23(4):345-356. doi: 10.1016/0304-3959(85)90004-1. PMID 4088697
- [Background] Cano A, Leonard MT, Franz A. The significant other version of the Pain Catastrophizing Scale (PCS-S): preliminary validation. Pain. 2005 Dec 15;119(1-3):26-37. doi: 10.1016/j.pain.2005.09.009. Epub 2005 Nov 17. PMID 16298062
- [Background] Kindt S, Vansteenkiste M, Loeys T, Cano A, Lauwerier E, Verhofstadt LL, Goubert L. When Is Helping your Partner with Chronic Pain a Burden? The Relation Between Helping Motivation and Personal and Relational Functioning. Pain Med. 2015 Sep;16(9):1732-44. doi: 10.1111/pme.12766. Epub 2015 Apr 30. PMID 25929153
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Leonard MT, Cano A, Johansen AB. Chronic pain in a couples context: a review and integration of theoretical models and empirical evidence. J Pain. 2006 Jun;7(6):377-90. doi: 10.1016/j.jpain.2006.01.442. PMID 16750794
- [Background] Martire LM, Stephens MA, Mogle J, Schulz R, Brach J, Keefe FJ. Daily spousal influence on physical activity in knee osteoarthritis. Ann Behav Med. 2013 Apr;45(2):213-23. doi: 10.1007/s12160-012-9442-x. PMID 23161472
- [Background] Uysal A, Ascigil E, Turunc G. Spousal autonomy support, need satisfaction, and well-being in individuals with chronic pain: A longitudinal study. J Behav Med. 2017 Apr;40(2):281-292. doi: 10.1007/s10865-016-9783-1. Epub 2016 Aug 19. PMID 27541643
- See also: Online form for individuals who would like to be contacted about participating in the study. — https://iitcop.az1.qualtrics.com/jfe/form/SV_eUHXgkcdRmHtNdj